CLINICAL TRIAL: NCT00765804
Title: Evaluation of Dexamethasone Phosphate Delivered by Ocular Iontophoresis for Treatment of Dry Eye in the Controlled Adverse Environment Model
Brief Title: Safety and Efficacy Study of Iontophoresis and Dexamethasone Phosphate to Treat Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Stephen From/Chief Executive Officer, Eyegate Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-437-002
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye; Iontophoresis; Ophthalmic Delivery
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose: DP 7.5 mA-min at 2.5 mA (Active Comparator): Ocular Iontophoresis with EGP-437 (dexamethasone phosphate ophthalmic solution 40 mg/mL) 7.5 mA-min at 2.5 mA
  Interventions: Drug: EGP-437 with EyeGate® II System
- High Dose: DP 10.5 mA-min at 3.5 mA (Active Comparator): Ocular Iontophoresis with EGP-437 (dexamethasone phosphate ophthalmic solution 40 mg/mL) 10.5 mA-min at 3.5 mA
  Interventions: Drug: EGP-437 with EyeGate® II System
- Placebo: 10.5 mA-min at 3.5 mA (Placebo Comparator): Ocular Iontophoresis with Placebo (sodium citrate buffer solution 100 mM at 10.5 mA-min at 3.5 mA)
  Interventions: Drug: Sodium citrate buffer solution with EyeGate® II System

INTERVENTIONS:
Drug: EGP-437 with EyeGate® II System — Transscleral iontophoretic delivery of EGP-437 (dexamethasone phosphate ophthalmic solution 40 mg/mL) delivered via EyeGate® II Drug Delivery System
  Other Names: Dexamethasone phosphate ophthalmic solution
  Arms: High Dose: DP 10.5 mA-min at 3.5 mA; Low Dose: DP 7.5 mA-min at 2.5 mA
Drug: Sodium citrate buffer solution with EyeGate® II System — Transscleral iontophoretic delivery of sodium citrate buffer solution 100 mM delivered via EyeGate® II Drug Delivery System
  Other Names: Sodium citrate buffer solution
  Arms: Placebo: 10.5 mA-min at 3.5 mA

SUMMARY:
The purpose of this study is to assess the safety and efficacy of iontophoretic delivery of dexamethasone phosphate ophthalmic solution using the EyeGate® II Drug Delivery System in patients with dry eye.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety and efficacy of Ocular Iontophoresis with Dexamethasone Phosphate 40 mg/mL 7.5 mA-min at 2.5 mA and Ocular Iontophoresis with Dexamethasone Phosphate 40 mg/mL 10.5 mA-min at 3.5 mA compared to placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Have a reported history of dry eye in each eye
* Be at least 12 years of age
* Demonstrate a response when exposed to the Controlled Adverse Environment model

Exclusion Criteria:

* Have contraindications to the use of the test articles
* Have known allergy or sensitivity to the study medication or their components (including corticosteroids)
* Have any ocular infections, active ocular inflammation or preauricular lymphadenopathy
* Be current contact lens wearers or wear contacts during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Sign: Corneal fluorescein staining after CAE exposure at Visit 5 | Visit 5 (Day 7 ± 2 Days)
  Corneal fluorescein staining after CAE exposure at Visit 5 as measured by the ORA scale.
Symptom: Ocular discomfort during CAE exposure at Visit 5 | Visit 5 (Day 7 ± 2 Days)
  Symptom: Ocular discomfort during CAE exposure at Visit 5 as measured by ORA scale.

SECONDARY OUTCOMES:
Sign: Fluorescein staining at each visit over 3 weeks | 7 visits / 3 weeks
  Fluorescein staining (each region) as measured by the ORA and NEI Scales at each of 7 visits over 3 weeks
Symptom: Ocular discomfort pre and post CAE | Visit 1 (Day -7 ± 2 Days), Visit 3 (Day 0), and Visit 5 (Day 7 ± 2 Days)
  Symptom: Ocular discomfort pre and post CAE (ORA Scale)at 3 visits (Visits 1, 3, and 5)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — ORA, Inc.
Locations (2):
- United States (2):
  - Ophthalmic Research Associates, Andover, Massachusetts
  - Ophthalmic Research Associates, North Andover, Massachusetts